CLINICAL TRIAL: NCT04656067
Title: Comparative Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate to Reduce Blood Loss Intraoperative and Post Operative During Elective Cesarean Section
Brief Title: Comparative Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Principal Investigator, DR.ABDELAZIM, Assistant specialist, Egymedicalpedia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR,ABDELAZIM SOBHI
Record Dates: First submitted 2020-11-26; First posted 2020-12-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-02

CONDITIONS: Blood Loss, Surgical; Blood Loss, Postoperative
Keywords: blood loss; Cesarean Section; Oxytocin; Tranexamic acid(Kapron); Etamsylate(Dicynon).
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage; Hemorrhage | interventions — Ethamsylate; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin(only) (Active Comparator): oxytocin is given IV infusion 5-10 minutes before the start of skin incision in the Elective Cesarean Section
  Interventions: Drug: Oxytocin ,Tranexamic acid and Ethamsylate
- Tranexamic acid and Ethamsylate (Active Comparator): Tranexamic acid and Ethamsylate are given IV slowly 5-10 minutes before the start of skin incision in the Elective Cesarean Section
  Interventions: Drug: Oxytocin ,Tranexamic acid and Ethamsylate

INTERVENTIONS:
Drug: Oxytocin ,Tranexamic acid and Ethamsylate — Is to compare blood loss during elective cesarean section intraoperative and postoperative in cases receiving Oxytocin versus Tranexamic acid and Ethamsylate
  Other Names: Syntocinon , Kapron; Dicynon

SUMMARY:
Comparative Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate, Pre-operative Administration.

DETAILED DESCRIPTION:
Caesarean Delivery commonly referred to as caesarean section and occasionally caesarean birth is defined as the delivery of a foetus(es) through surgical incisions made through the anterior abdominal wall (technically referred to as laparotomy) and the anterior uterine wall (technically denoted to as hysterotomy).

Obstetric Hemorrhage (Intra operative OR post operative bleeding)is still the major cause of maternal morbidity and mortality worldwide contributing to nearly 25% of direct maternal deaths. And accounts for 50% of maternal mortality in low-income countries.

So many Strategies reducing the intraoperative blood loss or post operative blood loss could be helpful in decreasing the risks of blood transfusion and the postoperative maternal morbidity.

So these Medications are such as Oxytocin, Carbetocin, Misoprostol, Prostaglandin F2 alpha, methylergonovine, Tranexamic acid and Etamsylate . have been tried before to control bleeding during and after Cesarean Section.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant females admitted for elective Cesarean Section.
2. Gestational age (38 to 41 weeks).
3. Age of the participants: 20 to 40 years.
4. Body Mass Index (18.5 - 29.9).
5. Singleton living fetus.
6. No medical disorders.
7. Informed written consent from the candidates.

Exclusion criteria:

1. - Medical and surgical disorders as thyroid dysfunction, which was excluded by routine thyroid function test (free T3, free T4, and thyroid-stimulating hormone(TSH), all of them should be within normal limits).
2. -Bleeding tendency, was excluded by platelet count, coagulation time, bleeding time, prothrombin time, partial thromboplastin time, and thrombin time (all should be within normal).
3. -Acute and chronic liver or kidney diseases; blood disorders, such as anemia.
4. -Allergy to Tranexamic acid or any drug used.
5. -Risk factors for PPH, such as polyhydramnios, fetal macrosomia, antepartum hemorrhage.
6. - Abnormal placentae such as placenta previa and placental abruption.
7. -Pregnancy complications such as severe pre-eclampsia, Gestational HTN, Gestational DM, and multi Fetal pregnancies, those requiring blood transfusion.
8. - Patients who refused spinal anesthesia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative and Post operative bleeding(defined as blood loss ≥500 cc) | First 2 hours after C-Section
  Outcome of the study will be measured in terms of assessment of Hemoglobin level and Hematocrit level pre and post operatively.

SECONDARY OUTCOMES:
Sever PPH as bleeding is >1000 cc | first 24 hours after C-Section
  Outcome of the study will be measured in terms of assessment of Hemoglobin level and Hematocrit level post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.,AbdelSattar M Farhan, Professor, Principal Investigator — Al-Azhar University, Faculty of medicine for boys; Dr.,ElSayed A. ElDesouky, Professor, Principal Investigator — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Sayed Galal Hospital and Shoubra General Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Is to compare blood loss during elective cesarean section intraoperative and postoperative in cases receiving Oxytocin versus Tranexamic acid and Etamsylate .